CLINICAL TRIAL: NCT03787628
Title: Cannabidiol Effects on Craving and Relapse Prevention in Opioid Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Edythe London, Distinguished Professor in Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-001748; 5UG3DA048388-03 (NIH)
Record Dates: First submitted 2018-12-17; First posted 2018-12-26 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Opioid-use Disorder
Keywords: Buprenorphine; Cannabidiol; Opioid Use disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (CBD) 600 mg (Active Comparator): Thirty participants who meet all eligibility criteria will be randomized to receive CBD (ATL5; Ananda Scientific) at a dose of 600 mg.
  Interventions: Drug: Cannabidiol (CBD) 600 mg
- Placebo (Placebo Comparator): Thirty participants who meet all eligibility criteria will be randomized to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol (CBD) 600 mg — CBD (300 mg) will be administered orally twice daily in the morning and again in the afternoon. The active ingredient in the Ananda investigational new drug, ATL5, is cannabidiol (CBD), extracted from hemp, at a 10% strength (softgel capsules with 100 mg/ml of CBD per capsule). The novel formulation is based on the principle that a water-free mixture of some concentrated inactive ingredients (excipients) self-assemble spontaneously into liquid nanodomains that contain the active component CBD. ATL5 Softgel Capsules will be manufactured by Baxco Pharmaceutical Inc. (California, USA) under cGMP conditions.
  Other Names: ATL5 (Ananda Scientific)
  Arms: Cannabidiol (CBD) 600 mg
Drug: Placebo — The placebo softgel capsule formulation will have a composition with the same relative proportions as the CBD ATL5 Softgel Capsules. This formulation will be manufactured by Baxco Pharmaceutical Inc. under cGMP conditions. The amount (number of softgel capsules) of placebo will be administered to match that of the active compound, daily in the morning and afternoon for each of 28 days.
  Other Names: Placebo for ATL5 (Ananda Ccientific)
  Arms: Placebo

SUMMARY:
This research aims to determine the effects and safety of cannabidiol (CBD) (ATL5 softgel capsules) as an adjunctive therapy for patients who have Opioid Use Disorder and are taking buprenorphine + naloxone or methadone. Buprenorphine + naloxone and methadone is an approved treatment for Opioid Use Disorder, but relapse to opioid misuse is common among patients who receive this treatment. Finding an adjunctive treatment for these patients would be helpful.

We will recruit participants from the Tarzana Treatment Center (TTC) in the San Fernando Valley. They will be receiving buprenorphine + naloxone or methadone as part of residential therapy. Potential participants who pass initial screening and wish to continue in the study will provide written, informed consent and will complete a 2-day evaluation, including blood and urine tests, questionnaires about their mood, medical, psychiatric and drug use history and physical exam.

Up to 60 participants who meet all eligibility criteria will be invited to complete baseline assessments (blood and urine tests, questionnaires), and will be assigned randomly to receive CBD (600 mg/day) or placebo, corresponding to two groups of up to 30 participants each.

After the baseline measurements, participants will take part in a 28-day treatment phase for 4 weeks. They will take the study medication under supervision (CBD 300 mg twice daily or placebo). Questionnaires on opioid craving, withdrawal, and mood symptoms will be administered daily during the treatment period, excluding weekends. After the 28-day intervention, participants will complete the questionnaires and undergo urine drug tests in 4 weekly follow-up visits.

The study will last ~10 weeks, comprising three periods: a screening period (2-weeks when participants are stabilized on buprenorphine + naloxone or methadone in residential treatment at the Tarzana Treatment Center), a treatment period (4 weeks when study CBD or placebo is administered at Tarzana Treatment Center), and a follow-up period (4 weeks after termination of the test intervention).

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo controlled, study of cannabidiol (CBD) (600 mg/day) as an adjunctive therapy to buprenorphine + naloxone or methadone in patients who have Opioid Use Disorder and are receiving residential behavioral therapy, including cognitive behavioral therapy. The primary endpoint will be safety and tolerability of CBD in these patients, as indicated by the incidence of treatment-emergent adverse events (n/% per group). Participants will be evaluated via measurement of cardiovascular parameters (heart rate, blood pressure, and cardiac rhythm and conduction on EKG), other vital signs, liver enzymes, pulse oximetry, adverse events, and pharmacokinetics. Secondary measures will include cue-induced craving, reductions in spontaneous craving, opioid withdrawal, and negative affective states.

Patients will be recruited from the Tarzana Treatment Center (TTC) in the San Fernando Valley, where buprenorphine + naloxone or methadone (as part of their treatment) and CBD (as part of this protocol) will be administered. Tarzana Treatment Centers, Inc. is a community-based, private non-profit behavioral healthcare organization located in Southern California with several agency sites, including the one in the San Fernando Valley, where this protocol will be conducted. TTC delivers drug and alcohol use treatment, has been accredited by the Joint Commission on Accreditation of Healthcare Organizations (JCAHO) since 1987, and has a workforce that includes physicians, psychologists, and nurses. TTC's substance use treatment approach includes residential programs that are overseen by a Program Director and are staffed by a clinical supervisor, operations supervisor, counselors, interns, nursing staff and 24/7 technicians. Groups and services include an education group, process group, 12-step, family group, mental health services and recreation skills. Cognitive-behavioral treatment is used in both individual and group therapy to address craving and relapse issues and in the treatment of mental health problems.

Up to 75 participants who meet all eligibility criteria will be invited to complete baseline assessments (blood and urine tests, questionnaires), and will be assigned randomly to receive CBD or placebo, corresponding to two groups of up to 30 participants each. Within each group, participants will be randomized by baseline buprenorphine plasma level (either below or ≥ 2 ng/ml).

The study will comprise three periods: 1) a screening period (~7-14-days) while participants are stabilized on buprenorphine + naloxone; 2) a 4-week treatment period when study medication will be administered; and 3) a 4-week follow-up period after termination of treatment with the study medication. Cue-induced craving sessions will be conducted at three times: Day 0 (baseline), Day 7 (when a steady state of CBD should have been reached; half-life of CBD after oral administration is 18-32 h), and Day 28 (end of treatment).

Adherence to medication in the trial will be assured as the participant will take the test medication (CBD or placebo) under supervision daily. Blood samples will be collected to determine plasma concentrations of CBD, buprenorphine, and laboratory assessments of safety. Cue-induced craving and other measures of craving and affect will be collected repeatedly during the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and speak English and has provided written informed consent.
* Age of 18-65 years (inclusive).
* Meeting criteria for an OUD according to the MINI for ≥ 3 months before screening.
* Self-report of opioid use in the 60 days before screening; verified by treatment center records.
* On a stable dose of ≥12 mg buprenorphine, either alone, or in combination with naloxone (buprenorphine/naloxone ratio of 4/1) for at least 7 days prior to starting and for the duration of the treatment phase of the study. OR, receiving methadone maintenance therapy for at least 7 days prior to starting and for the duration of the treatment phase of the study.
* If female, being surgically sterile or willing to use birth control (e.g., oral contraceptives, condoms, intrauterine device) or willingness to abstain from sex throughout the study.
* Body Mass Index (BMI) between 17.5 and 35 kg/m2; total body weight > 110 lb (50 kg).
* Currently in residential treatment at the Tarzana Treatment Center.

Exclusion Criteria:

* History of sensitivity to a CBD product or any of the ingredients in the study drug, including glycerin or gelatin.
* A condition that may affect drug absorption (e.g., gastrectomy).
* Taking a medications that has clinically significant interactions with CBD or are contraindicated for the study (check with study physician).
* Positive urine test for THC at screening.
* Self-report of using CBD at screening.
* PK analysis at screening showing evidence of CBD use (a signal that is ≥ three times the background noise at the corresponding CBD retention time and MS2 transition).
* Physiological dependence on alcohol or a sedative-hypnotic benzodiazepine drug.
* Current medication-assisted treatment with naltrexone.
* Acute opioid withdrawal symptoms, as defined by a score on the COWS > 4.
* Clinical laboratory finding of AST or ALT > 3 times the upper limit of normal (ULN) or bilirubin > 1.5 times ULN.
* AIDS or HIV positive status (because treatment medications have potential interactions with CBD).
* Pregnancy or lactation.
* Clinically significant EKG abnormalities, as determined by the study physician, including the following: QTc >450 msec (men) or >470 (women) or QRS interval >120 msec (If QTc or QRS interval exceed these cutoff points, EKG will be repeated twice and the average of the three QTc values used to determine eligibility.), congenital long QT syndrome, history of prolonged QT in the 3 months before screening, corrected QT interval (Fridericia's - QTcF) >450 msec (male) or >470 msec (female) or history of risk factors for Torsades de Pointes.
* For women: any value outside reference ranges on a hormonal battery [estradiol, follicle-stimulating hormone, free thyroxine index, luteinizing hormone, prolactin, T3 uptake, thyroid-stimulating hormone, and thyroxine], followed by an abnormal ovarian ultrasound finding.
* Clinically significant cardiovascular, hematologic, hepatic, renal, or endocrine abnormalities, as determined by the study physician.
* Meeting criteria on the MINI for schizophrenia, Bipolar I disorder, psychotic disorder, having active suicidal ideation, or suicide attempt in the past 12 months. Or, answers "yes" to questions 4 or 5 on C-SSRS. NOTE: Participants with other psychiatric conditions, such as major depression, generalized anxiety, dysthymia, social phobia or specific phobia may be enrolled in the study if they are clinically stable.
* On the cue-induced opiate craving task at screening, the participant does not have a score of at least 25 (on a visual analogue scale with a maximum score of 100) for at least one image within one category. Note: Groups of images may be separated into smoking cues, pills and bottles, and injection paraphernalia. For example, for injection cues, a picture of a needle and syringe may elicit a craving response, though other images in the same group (i.e., picture of arm with vein bulging) do not elicit craving.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edythe London, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Tarzana Treatment Centers, Tarzana, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was from May 19, 2022 through March 12, 2024. Recruitment was at the Tarzana Treatment Center (TTC), where buprenorphine (as part of their treatment) and CBD (as part of this protocol) were administered. Of 35 enrolled participants, 30 started the study and received CBD or placebo (3 withdrew consent before treatment, 1 was disqualified because opioid use was outside the acceptable window, and 1 was nonmedically discharged prior to receiving the first dose).
Pre-assignment Details: Of 170 participants pre-screened, 97 were ineligible. Seventy-one were screened. Of these, 36 were excluded, 35 were enrolled, and 30 started the study and received at least one dose of medication (Safety Population).
Groups:
- Cannabidiol (CBD) 600 mg: Participants who eligibility criteria were be randomized to receive CBD (ATL5; Ananda Scientific) at a dose of 600 mg.
  Cannabidiol (CBD) 600 mg: CBD (300 mg) was administered orally twice daily in the morning and again in the afternoon. The active ingredient in the Ananda investigational new drug, ATL5, is cannabidiol (CBD), extracted from hemp, at a 10% strength (softgel capsules with 100 mg/ml of CBD per capsule). The novel formulation is based on the principle that a water-free mixture of some concentrated inactive ingredients (excipients) self-assemble spontaneously into liquid nanodomains that contain the active component CBD. ATL5 Softgel Capsules was manufactured by Baxco Pharmaceutical Inc. (California, USA) under cGMP conditions.
- Placebo: Up to 30 participants who meet all eligibility criteria were randomized to receive placebo.
  Placebo: The placebo softgel capsule formulation had a composition with the same relative proportions as the CBD ATL5 Softgel Capsules. This formulation was manufactured by Baxco Pharmaceutical Inc. under cGMP conditions. The amount (number of softgel capsules) of placebo was administered to match that of the active compound, daily in the morning and afternoon for each of 28 days.
Period: Overall Study
Arm/Group | Cannabidiol (CBD) 600 mg | Placebo
Started | 18 | 12
Completed | 11 | 6
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Cannabidiol (CBD) 600 mg: Up to 30 participants who meet all eligibility criteria will be randomized to receive CBD (ATL5; Ananda Scientific) at a dose of 600 mg.
- Placebo: Up to 30 participants who meet all eligibility criteria will be randomized to receive placebo.
- Total: Total of all reporting groups
Arm/Group | Cannabidiol (CBD) 600 mg | Placebo | Total
Number analyzed (Participants) | 18 | 12 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (11.34) | 35.0 (7.98) | 36.1 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 13 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 0 | 1 | 1
  White | 16 | 10 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint Will be Safety and Tolerability of CBD.
Description: Number of participants with treatment-emergent adverse events (n/% per treatment group).
Time Frame: Days 1-56
Population: The population reported on is the Safety Population, which received at least one dose of active medication or placebo.
Measure: Number; unit: participants
Groups:
- CBD 600 mg: This group reeived the active treatment, CBD at a dose of 600 mg/day.
- Placebo: This group received a placebo that was identical in number and appearance of capsules that contained CBD. The excipients in the active formulation were included here.
Arm/Group | CBD 600 mg | Placebo
Number analyzed (Participants) | 18 | 12
participants | 13 | 4

2. Secondary Outcome: The Extent to Which CBD Reduces Cue-induced Craving for Opioids.
Description: Cue-induced craving was measured at baseline, Day 7, and Day 28, when participants completed a cue-induced craving task in which they viewed pictures of neutral and opioid-related cues and rated their level of opioid craving on an abbreviated (7-item) version of the Desire for Drug Questionnaire (DDQ). The DDQ is comprised of Likert-style responses ranging from 1 (strongly disagree) to 7 (strongly agree), with total scores on the 7-item scale ranging from 7 to 49, with higher scores reflecting higher craving. The measure of cue-induced craving was derived by subtracting DDQ scores following neutral cues from DDQ scores following opioid cues (range = -42 to 42), with higher scores reflecting greater craving following opioid cues than neutral cues.
Time Frame: Before dosing on Day 0 (baseline without CBD) and on Days 7 and 28 after treatment with CBD. The group means below reflect the overall group means across time points as reported from descriptive statistics in the Generalized Linear Mixed Model (GLMM).
Population: The analysis populaton was the Safety Population (participants who received at least one dose of test compound).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol (CBD) 600 mg | Placebo
Number analyzed (Participants) | 18 | 12
score on a scale | 4.45 (6.54) | 7.19 (6.85)
Statistical Analysis 1: Comparison: Cannabidiol (CBD) 600 mg vs Placebo; Test type: Other — Generalized linear mixed model (GLMM) testing the main effect of group and time, and the group X time interaction; p = 0.41, Mixed Models Analysis — P-value reflects the test of the interaction between group and time on the measure of cue-induced craving; F-test = 0.703 — Estimated value reflects the f test of the interaction between group and time on the measure of cue-induced craving (degrees of freedom = 1, 67)

3. Other Pre Specified Outcome: Spontaneous Opioid Craving Using the Penn Alcohol Craving Scale (PACS), Adapted for Opioid Craving.
Description: The Penn Alcohol Craving Scale (PACS) is a brief 4-item self-report measure of spontaneous alcohol craving. In the current study, the items were adapted to measure opioid craving instead of alcohol craving. Responses pertain to opioid craving in the last 24 hours and are measured on a Likert-scale (ranging from 0 to 6), with total scores ranging from 0 to 24. Higher total scores indicate higher levels of spontaneous opioid craving.
Time Frame: Before dosing (Day 0), daily during treatment period (28 days), and weekly during follow-up (up to 4 weeks). Group means below reflect overall group means across time points as reported from descriptive statistics in the Generalized Linear Mixed Model.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBD 600 mg | Placebo
Number analyzed (Participants) | 18 | 12
score on a scale | 5.11 (3.97) | 5.62 (4.48)
Statistical Analysis 1: Comparison: CBD 600 mg vs Placebo; Test type: Other — Generalized linear mixed model (GLMM) testing the main effect of group and time, and the group X time interaction; p = 0.99, Mixed Models Analysis — P-value reflects the test of the interaction between group and time on the measure of spontaneous craving; F-test = 0.00 — Estimated value reflects the f test of the interaction between group and time on spontaneous craving (degrees of freedom = 1, 550)

4. Other Pre Specified Outcome: State Anxiety Subscale of the Spielberger State-Trait Anxiety Inventory (STAI).
Description: State anxiety is assessed with the 20-item self-report subscale from the 40-item Spielberger State-Trait Anxiety Inventory (STAI). The state anxiety subscale evaluates how respondents feel "now", in the present moment. All items are rated on a Likert scale from 1 ("not at all") to 4 ("very much so"), with total scores on the state anxiety subscale ranging from 20 to 80. Higher total scores indicate greater state anxiety.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBD 600 mg | Placebo
Number analyzed (Participants) | 18 | 12
score on a scale | 33.25 (11.18) | 36.25 (8.17)
Statistical Analysis 1: Comparison: CBD 600 mg vs Placebo; Test type: Other — Generalized linear mixed model (GLMM) testing the main effect of group and time, and the group X time interaction; p = 0.84, Mixed Models Analysis — P-value reflects the test of the interaction between group and time on the measure of state anxiety; F-test = 0.04 — Estimated value reflects the f test of the interaction between group and time on state anxiety (degrees of freedom = 1, 550)

5. Other Pre Specified Outcome: Negative Affect Subscale From the Positive and Negative Affect Schedule (PANAS).
Description: Negative affect is assessed using the 15-item negative affect subscale from the 30-item Positive and Negative Affect Schedule (PANAS). Each item is rated on a 5-point scale ranging from 1 (not at all) to 5 (extremely), with total scores on the negative affect subscale ranging from 15 to 75. Higher scores reflect greater negative affect.
Time Frame: Before dosing (Day 0), daily during treatment period (28 days), and weekly during follow-up (up to 4 weeks). Group means reflect overall group means across time points as reported from descriptive statistics in the Generalized Linear Mixed Model.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBD 600 mg | Placebo
Number analyzed (Participants) | 18 | 12
score on a scale | 18.97 (6.70) | 19.15 (5.48)
Statistical Analysis 1: Comparison: CBD 600 mg vs Placebo; Test type: Other — Generalized linear mixed model (GLMM) testing the main effect of group and time, and the group X time interaction; p = 0.60, Mixed Models Analysis — P-value reflects the test of the interaction between group and time on the measure of negative affect; F-test = 0.27 — Estimated value reflects the f test of the interaction between group and time on negative affect (degrees of freedom = 1, 550)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded over a 28-day treatment perioid and in follow-up sessions through Day 56.
Description: Adverse Events, obtained in self-reports, were recorded dalily.
  Lab tests and procedures also were performed to monitor safety. Assessment times were during baseline, the treatment period (28 days) and follow up (up to 56 days from the start of treatment):
  1. Comprehensive metabolic panel (key tests: AST, ALT, INR)
  2. Assessment of Sedation (Observed Observer's Assessment of Alertness/Sedation Scale, pulse oximetry)
  3. Electrocardiogram
  4. Ovarian hormone battery (females)
Arm/Group | Cannabidiol (CBD) 600 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 8/18 | 3/12
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/12
Other Adverse Events (participants affected / at risk) | 8/18 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cannabidiol (CBD) 600 mg (N=18) | Placebo (N=12)
Liver function test (Investigations) | 1 (1) | 0 (0) — abnormal LFTs
abdominal pain/abdominal cramps or Nausea or Constipation (Gastrointestinal disorders) | 6 (7) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Oxygen saturaton decreased (Investigations) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT03787628/Prot_002.pdf
  • Statistical Analysis Plan (2024-08-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT03787628/SAP_001.pdf